CLINICAL TRIAL: NCT02132767
Title: Rate Control Versus Rhythm Control For Postoperative Atrial Fibrillation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Annetine Gelijns, Professor and Chair, Health Evidence and Policy, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 08-1078-00007; 5U01HL088942-08 (NIH)
Record Dates: First submitted 2014-05-05; First posted 2014-05-07 (Estimated); Results first posted 2017-01-18 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2019-02

CONDITIONS: Postoperative Atrial Fibrillation
Keywords: Heart surgery; Cardiac surgery; Coronary artery bypass; Mitral valve surgery; Aortic valve surgery; Atrial fibrillation; Atrial flutter; Cardiac arrhythmia; Valve surgery
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter; Arrhythmias, Cardiac | interventions — Amiodarone; Electric Countershock; Heart Rate; Adrenergic beta-Antagonists; Calcium Channel Blockers; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rhythm control (Active Comparator): Rhythm Control in post-operative AF
  Amiodarone and/or DC-cardioversion
  Amiodarone Initial Dose
  * Oral: 400 mg po TID for 3 days is recommended
  * For patients incapable of taking oral: 150 mg IV bolus over 10 min, then 1 mg/min over 6 hours followed by 0.5 mg/min over 18 hours Maintenance Dose
  * Oral: at least 200 mg/day to be continued until 60 days after randomization
  * If drug cannot be given orally or via NG tube: 0.5 mg/min administered through central line (e.g., PICC) until oral dosing is started
  DC-Cardioversion - frequency and duration determined by medical professional as medically needed
  Interventions: Drug: Amiodarone; Procedure: DC-cardioversion
- Rate control (Active Comparator): Rate Control in post-operative AF
  Beta-blocker and/or Calcium channel blockers and/or Digoxin
  Dose, frequency and duration determined by medical professional as medically needed
  Interventions: Drug: Rate Control

INTERVENTIONS:
Drug: Amiodarone — Amiodarone Initial Dose
  * Oral: 400 mg po TID for 3 days is recommended
  * For patients incapable of taking oral: 150 mg IV bolus over 10 min, then 1 mg/min over 6 hours followed by 0.5 mg/min over 18 hours Maintenance Dose
  * Oral: at least 200 mg/day to be continued until 60 days after randomization
  * If drug cannot be given orally or via NG tube: 0.5 mg/min administered through central line (e.g., PICC) until oral dosing is started
  Other Names: Cordarone
  Arms: Rhythm control
Procedure: DC-cardioversion — DC-Cardioversion - frequency and duration determined by medical professional as medically needed
  Other Names: Direct Current Cardioversion
  Arms: Rhythm control
Drug: Rate Control — Beta-blocker and/or Calcium channel blockers and/or Digoxin - Dose, frequency and duration determined by medical professional as medically needed
  Other Names: Beta-blocker; Calcium channel blockers; Digoxin
  Arms: Rate control

SUMMARY:
The purpose of this study is to compare the therapeutic strategies of rate control versus rhythm control in cardiac surgery patients who develop in-hospital postoperative atrial fibrillation or atrial flutter (AF). In patients who develop AF during hospitalization after cardiac surgery, the hypothesis is that a strategy of rhythm control will reduce days in hospital within 60 days of the occurrence of AF compared to a strategy of rate control.

DETAILED DESCRIPTION:
The purpose of the research is to compare two strategies for treating atrial fibrillation or atrial flutter, both of which are referred to as AF, after cardiac surgery. AF is the most common complication after cardiac surgery. AF is when the upper chambers of the heart (atria) experience disorganized electrical activity which causes the heart beat to be irregular. The two treatment strategies to be used in this study are called rhythm control and rate control. The rhythm control strategy will attempt to bring the heart beat back to a regular rhythm using treatments known and approved to control heart rhythm. The rate control strategy will attempt to bring the heart rate to less than 100 beats per minute at rest using medications known and recommended to control heart rate. Both strategies are commonly used to treat AF. All of the medications that will be used in this study are the standard of care for use in patients experiencing AF. This research seeks to determine whether rhythm control is better than rate control in patients with AF after cardiac surgery.

ELIGIBILITY:
Enrollment Inclusion Criteria:

* Age > 18 years
* Undergoing heart surgery for coronary artery bypass (on-pump or off-pump CABG) and/or valve repair or replacement (excluding mechanical valves), including re-operations
* Hemodynamically stable

Randomization Inclusion Criteria

* AF that persists for > 60 minutes or recurrent (more than one) episodes of AF up to 7 days after surgery during the index hospitalization.

Exclusion Criteria:

* LVAD insertion or heart transplantation
* Maze procedure
* TAVR
* History of or planned mechanical valve replacement
* Correction of complex congenital cardiac defect (excluding bicuspid aortic valve, atrial septal defect or PFO)
* History of AF or AFL
* History of AF or AFL ablation
* Contraindications to warfarin or amiodarone
* Need for long-term anticoagulation
* Concurrent participation in an interventional (drug or device) trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 523 (Actual)
Dates: Start 2014-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Wiesel, MD, Study Chair — Cardiothoracic Surgical Trials Network; Patrick T O'Gara, MD, Study Chair — Cardiothoracic Surgical Trials Network
Locations (23):
- United States (17):
  - University of Southern California, Los Angeles, California
  - Emory University, Atlanta, Georgia
  - University of Maryland, Baltimore, Maryland
  - NIH Heart Center at Suburban Hospital, Bethesda, Maryland
  - University of Michigan Health Services, Ann Arbor, Michigan
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - Montefiore Einstein Heart Center, The Bronx, New York
  - Mission Hospital, Asheville, North Carolina
  - Duke University, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Baylor Research Institute, Plano, Texas
  - University of Virginia Health Systems, Charlottesville, Virginia
  - University of Wisconsin, Madison, Wisconsin
- Canada (6):
  - University of Alberta Hospital, Edmonton, Alberta
  - Toronto General Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
  - Hôpital du Sacré-Cœur de Montréal, Montreal, Quebec
  - Institut Universitaire de Cardiologie de Quebec (Hopital Laval), Québec, Quebec

REFERENCES:
- [Derived] Afifi A. CTS trials network: Rate control vs rhythm control for atrial fibrillation after cardiac surgery - Do bitter pills have blessed effects? Glob Cardiol Sci Pract. 2016 Jun 30;2016(2):e201615. doi: 10.21542/gcsp.2016.15. PMID 29043263
- [Derived] Gillinov AM, Bagiella E, Moskowitz AJ, Raiten JM, Groh MA, Bowdish ME, Ailawadi G, Kirkwood KA, Perrault LP, Parides MK, Smith RL 2nd, Kern JA, Dussault G, Hackmann AE, Jeffries NO, Miller MA, Taddei-Peters WC, Rose EA, Weisel RD, Williams DL, Mangusan RF, Argenziano M, Moquete EG, O'Sullivan KL, Pellerin M, Shah KJ, Gammie JS, Mayer ML, Voisine P, Gelijns AC, O'Gara PT, Mack MJ; CTSN. Rate Control versus Rhythm Control for Atrial Fibrillation after Cardiac Surgery. N Engl J Med. 2016 May 19;374(20):1911-21. doi: 10.1056/NEJMoa1602002. Epub 2016 Apr 4. PMID 27043047
- See also: Cardiothoracic Surgical Trials Network Website — http://www.ctsurgerynet.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Rate Control: Patients randomized to this arm will be treated with an initial strategy of rate control. The target heart rate is < 100 beats per minute at rest. The treating clinician will choose agents from the list of rate control medications below and employ these medications (singly or in combination) to achieve rate control. A patient who presents with AF and slow ventricular response rate (<60 beats per minute) may still be randomized to the rate control strategy; in such instances, rate control agents may be withheld or administered in low doses. Dose ranges, as defined in guidelines, for each of the rate control agents need to be adhered to. Simultaneous use of more than one of the categories of rate control agents should be done with caution due to risk of bradycardia.
  Rate Control Agents:
  Beta blockers (e.g. metoprolol, atenolol, carvedilol, esmolol) Calcium channel blockers (nondihydropyridine) (e.g. diltiazem, verapamil) Digoxin
- Rhythm Control: Patients assigned to an initial strategy of rhythm control will be treated with amiodarone alone or amiodarone plus direct current (DC) cardioversion if amiodarone alone does not eliminate AF within 48 hours. For patients who are hemodynamically stable but remain in AF, at least 24 hours of amiodarone should be administered before cardioversion is attempted. Cardioversion should be attempted, if possible, prior to the 48 hour duration to avoid the need for a TEE guided approach.
  If AF has been present for ≥ 48 hours and the patient has not been therapeutically anticoagulated, cardioversion should be TEE guided. When deemed to be clinically appropriate, patients in the rhythm control arm may also be treated with a rate control medication (e.g. beta blocker). In particular, a rate control medication may be indicated at the onset of AF.
Period: Overall Study
Arm/Group | Rate Control | Rhythm Control
Started | 262 | 261
Completed | 245 | 246
Not Completed | 17 | 15
Not completed — Death | 3 | 2
Not completed — Withdrawal by Subject | 10 | 9
Not completed — Lost to Follow-up | 4 | 4

BASELINE CHARACTERISTICS:
Population: All randomized patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Rate Control | Rhythm Control | Total
Number analyzed (Participants) | 262 | 261 | 523
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (9.8) | 68.4 (8.4) | 68.8 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 62 | 127
  Male | 197 | 199 | 396
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 12 | 22
  Not Hispanic or Latino | 252 | 249 | 501
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 13 | 3 | 16
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 5 | 5 | 10
  White | 242 | 250 | 492
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 32 | 29 | 61
  United States | 230 | 232 | 462

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Days in Hospital
Description: The total number of days in hospital for any hospitalization that occurs within 60 days of randomization to AF treatment strategy.
Time Frame: Within 60 days of randomization
Population: All randomized patients (intent to treat)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Rate Control | Rhythm Control
Number analyzed (Participants) | 262 | 261
days | 5.1 [3.0 to 7.4] | 5.0 [3.2 to 7.5]
Statistical Analysis 1: Comparison: Rate Control vs Rhythm Control; Test type: Superiority or Other; p = 0.76, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Time to Conversion to Sustained, Stable Non-AF Rhythm
Time Frame: Up to index hospital discharge or 7 days post surgery, whichever came first
Population: All randomized patients (intent to treat)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Rate Control | Rhythm Control
Number analyzed (Participants) | 262 | 261
days | 1.85 [0.46 to 4.81] | 0.95 [0.27 to 3.21]
Statistical Analysis 1: Comparison: Rate Control vs Rhythm Control; Test type: Superiority or Other; p = 0.003, Log Rank

3. Secondary Outcome: Heart Rhythm Comparison
Description: Compare heart rhythm (number of patients in sustained, stable non-AF rhythm) between treatment arms at hospital discharge
Time Frame: Hospital discharge
Measure: Number; unit: participants
Arm/Group | Rate Control | Rhythm Control
Number analyzed (Participants) | 257 | 261
participants | 231 | 244
Statistical Analysis 1: Comparison: Rate Control vs Rhythm Control; Test type: Superiority or Other; p = 0.14, Chi-squared

4. Secondary Outcome: Heart Rhythm Comparison
Description: Compare heart rhythm (patients in sustained, stable non-AF rhythm) between treatment arms at 30 days after randomization
Time Frame: 30 days after randomization
Measure: Number; unit: participants
Arm/Group | Rate Control | Rhythm Control
Number analyzed (Participants) | 242 | 248
participants | 220 | 223
Statistical Analysis 1: Comparison: Rate Control vs Rhythm Control; Test type: Superiority or Other; p = 0.71, Chi-squared

5. Secondary Outcome: Heart Rhythm Comparison
Description: Compare heart rhythm (number of patients in sustained, stable non-AF rhythm) between treatment arms at 60 days after randomization
Time Frame: 60 days after randomization
Measure: Number; unit: participants
Arm/Group | Rate Control | Rhythm Control
Number analyzed (Participants) | 234 | 236
participants | 220 | 231
Statistical Analysis 1: Comparison: Rate Control vs Rhythm Control; Test type: Superiority or Other; p = 0.03, Chi-squared

6. Secondary Outcome: Length of Stay (Index Hospitalization)
Description: Overall length of stay for the index hospitalization
Time Frame: Within 60 days post surgery
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Rate Control | Rhythm Control
Number analyzed (Participants) | 262 | 261
days | 4.3 [2.9 to 6.6] | 4.3 [3.0 to 7.0]
Statistical Analysis 1: Comparison: Rate Control vs Rhythm Control; Test type: Superiority or Other; p = 0.88, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Length of Stay (Rehospitalization, Including ED Visits)
Description: Compare length of stay between groups for any cause and AF-related hospitalizations, including ED visits
Time Frame: Within 60 days of randomization
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Rate Control | Rhythm Control
Number analyzed (Participants) | 262 | 261
days | 2.2 [0.6 to 5.0] | 2.1 [1.0 to 4.7]
Statistical Analysis 1: Comparison: Rate Control vs Rhythm Control; Test type: Superiority or Other; p = 0.82, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Outpatient Interventions
Description: Compare frequency of outpatient visits between groups for any cause and AF-related causes
Time Frame: Within 60 days of randomization
Measure: Number; unit: hospital stays < 24 hours
Arm/Group | Rate Control | Rhythm Control
Number analyzed (Participants) | 262 | 261
hospital stays < 24 hours | 5 | 4
Statistical Analysis 1: Comparison: Rate Control vs Rhythm Control; Test type: Superiority or Other; p = 0.73, Regression, Poisson

9. Secondary Outcome: AF- or Treatment-related Events
Time Frame: Within 60 days of randomization
Reporting Status: Not Posted

10. Secondary Outcome: Cost (Hospital)
Description: Compare cost of index hospitalization and cost of rehospitalizations (including ED visits) between groups
Time Frame: Within 60 days of randomization
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Rate Control | Rhythm Control
Serious Adverse Events (participants affected / at risk) | 71/262 | 73/261
Other Adverse Events (participants affected / at risk) | 29/262 | 26/261
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rate Control (N=262) | Rhythm Control (N=261)
Bleeding (General disorders) | 10 (11) | 6 (6)
Cardiac Arrhythmias (Cardiac disorders) | 20 (21) | 19 (23)
Cerebrovascular Thromboembolism (Nervous system disorders) | 4 (4) | 2 (2)
Heart Failure (Cardiac disorders) | 8 (9) | 7 (9)
Major Infection (Infections and infestations) | 23 (28) | 16 (22)
Non-Cerebral Thromboembolism (Vascular disorders) | 2 (2) | 0 (0)
Pericardial Fluid Collection (Cardiac disorders) | 2 (2) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 19 (23)
Renal Events (Renal and urinary disorders) | 5 (5) | 5 (6)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (8)
Anemia (General disorders) | 0 (0) | 3 (3)
Coumadin Toxicity (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hypotension/Syncope (Cardiac disorders) | 5 (6) | 3 (4)
Amiodarone Toxicity (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Abdominal Distress (Gastrointestinal disorders) | 2 (2) | 0 (0)
Chest Pain (Cardiac disorders) | 2 (2) | 5 (5)
Dysphagia (General disorders) | 0 (0) | 1 (1)
Fall Not Related to Syncope (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Heparin-Induced Thrombocytopenia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyperkalemia (General disorders) | 0 (0) | 1 (1)
Hypoglycemia (General disorders) | 1 (1) | 0 (0)
Ischemic Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nosocomial Fever (General disorders) | 0 (0) | 1 (1)
Peripheral Arterial Thrombus (Vascular disorders) | 0 (0) | 1 (1)
Peripheral Vascular Disease (Vascular disorders) | 0 (0) | 1 (1)
Peripheral Neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Right Groin Hematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sternal Wound Dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Encephalopathy (General disorders) | 1 (1) | 1 (1)
Post-Pericardiotomy Syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Small Bowel Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Non-Cerebral Thromboembolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rate Control (N=262) | Rhythm Control (N=261)
Bleeding (General disorders) | 2 (2) | 1 (2)
Cardiac Arrhythmias (Cardiac disorders) | 2 (2) | 7 (8)
Major infection (Infections and infestations) | 17 (18) | 11 (11)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Renal events (Renal and urinary disorders) | 3 (4) | 6 (6)
Superficial venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis left limb (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No